CLINICAL TRIAL: NCT02304094
Title: A Randomised Controlled Trial to Compare the Clinical Effectiveness of Lower Extremity Manipulation to That of Steroid Injection in the Treatment of Morton's Neuroma
Brief Title: Morton's Neuroma: Manipulation Versus Steroid Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Margaret University (Other)
Responsible Party: Principal Investigator, David Cashley, Mr David Cashley, Queen Margaret University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PDN001
Record Dates: First submitted 2014-11-24; First posted 2014-12-01 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Neuroma, Human Forefoot
MeSH Terms: conditions — Neuroma | interventions — Methylprednisolone; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- manipulation (Experimental): Those in the manipulation group shall have the lesser MTPJs of the affected foot manually manipulated using a high velocity, low amplitude thrust technique. They will be asked to return once each week for a further five weeks. At each visit the VAS and PTM measurements shall be repeated, as will the manual manipulation. They shall also be asked to return for a review in the sixth week.
  Interventions: Other: Manual manipulation
- Steroid (Active Comparator): Those randomised to the steroid group shall receive a single injection of 1 mL methylprednisolone [40 mg] and 1 mL 2% lignocaine. They shall then be asked to return for review in six weeks. A second injection may be offered at this point if clinically indicated.
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Drug: methylprednisolone — the steroid group shall receive a single injection of 1 mL methylprednisolone [40 mg] and 1 mL 2% lignocaine
  Arms: Steroid
Other: Manual manipulation — the manipulation group shall have the lesser MTPJs of the affected foot manually manipulated using a high velocity, low amplitude thrust technique
  Arms: manipulation

SUMMARY:
The aim of this study is to establish which of two treatment options is the preferred intervention in the treatment of Morton's Neuroma.

A randomised controlled trial shall be performed. Steroid injection is the current gold standard conservative treatment for this condition. Therefore, manipulation shall be compared to a control group receiving a steroid injection in an equality randomised controlled trial.

Outcomes will be compared using visual analogue pain scales (VAS), The Manchester-Oxford Foot Questionnaire (MOXFQ), The Foot and Ankle Ability Measure (FAAM), the SF-36 quality of life questionnaire and algometric pressure threshold testing. An improvement in either groups' VAS of 20mm above the other group shall be considered as the minimum worthwhile change as this has been identified as the minimum clinically important difference in pain between treatment groups in visual analogue pain scales.

There is limited research evidence to support the management of Morton's neuroma with steroid injection although its efficacy has only been demonstrated in the short term.

DETAILED DESCRIPTION:
Proposed Randomised Single Blind Study Aims and objectives The aim of this study is to establish which of two treatment options is the preferred intervention in the treatment of Morton's Neuroma.

Objectives. A systematic review of the literature shall be undertaken in order to inform the researchers. The Pressure Threshold Meter shall be validated for use in the foot.

A randomised controlled trial shall be performed. Steroid injection is the current gold standard conservative treatment for this condition. Therefore, manipulation shall be compared to a control group receiving a steroid injection in an equality randomised controlled trial.

Outcomes will be compared using visual analogue pain scales (VAS), The Manchester-Oxford Foot Questionnaire (MOXFQ), The Foot and Ankle Ability Measure (FAAM), the SF-36 quality of life questionnaire and algometric pressure threshold testing.

An improvement in either group VAS of 20mm above the other group shall be considered as the minimum worthwhile change as this has been identified as the minimum clinically important difference in pain between treatment groups in visual analogue pain scales (Thomson et al. 2013). The primary question will ask whether manipulation is beneficial in the treatment of MN. Secondary questions will be addressed, including, are the benefits of manipulation for Morton's neuroma long lasting, and do they out-perform the current conservative interventions at three months, six months and one year. Is PTM an accurate and reliable measurement tool for foot pain? Furthermore, does manipulation result in changes to mechanical loading during gait as seen on high resolution walkway analysis?

Ethics The main ethical issue is in asking subjects in pain to accept an experimental treatment.

The study has been designed in such a way as to ensure that no volunteers are denied treatment. There will also be an opportunity for those who have not benefited from their allocated treatment to receive the alternative treatment or another treatment entirely. Each volunteer shall have access to the standard treatment pathway at any time, should they wish to avail themselves of it. This shall be fully explained to all volunteers prior to enrolment in the study. At the completion of the study, all subjects shall have the treatment with the strongest outcome scores made available to them.

Patient Recruitment All patients from The Edinburgh foot and ankle surgical unit, QMU musculoskeletal clinic, Dundee Podiatry Clinic and from The Queen Margaret Hospital, Dunfermline with a suspicion of Morton's neuroma shall be invited to participate in the study. A member of the patient's existing clinical care team shall check whether they meet the study inclusion and exclusion criteria and make the initial approach to invite them to become involved with the study. They will also give the patient the participant information literature. Their active involvement in the study should amount to no more than the initial six weeks followed by review appointments at six weeks, then three, six, nine and twelve months.

Methods

1. Prior to the study, the pressure algometer, the ultrasound machine and the high resolution walkway will all be calibrated and validated.
2. Patients will be recruited from a variety of sources including Edinburgh Royal Infirmary, QMU, Margaret Rose Hospital, Dunfermline and The Dundee Podiatry Clinic.
3. The clinicians at the above sources shall identify potential subjects and assess them against the study's inclusion and exclusion criteria. Those who express an interest will be given the written information in the form of a patient information sheet [appendix 1] which describes the study in detail. They will then be invited to contact the chief investigator (David Cashley) should they choose to become involved.
4. Detailed information about the study will be given by the chief investigator to each potential subject who makes contact and they will then be given an appointment for the QMU gait analysis laboratory. There will be a minimum three month wash-out period for all subjects who have previously had any treatment for Morton's neuroma.
5. Those who attend QMU will be invited to ask questions about the study and raise any concerns that they may have. They will then be asked if they still want to participate in the study. If they agree, they will be asked to sign a consent form [appendix 2] and will have a study participation number allocated to them at this point in order to aide anonymous data collection. The chief investigator will then gather further information to include age, gender, duration and location of symptoms.
6. Participants who no longer wish to be involved in the study will be directed into the Musculoskeletal clinic at QMU for further assessment and treatment.
7. A baseline set of VAS [appendix 3] and QoL [appendix 4] scores will then be completed by all participants. All VAS and QoL questionnaires will be completed solely by the subject, with no intervention from any third party. This will serve to blind the researcher to the VAS and questionnaire measurements until the study is complete.
8. The following clinical tests shall be performed on all participants in a predetermined order that changes for each participant in order to limit the effect of hyperalgesia (from repetitive testing) adversely affecting any single test. The tests are as follows; Lateral squeeze test; Digital nerve stretch test; Gauthier's test; Sullivan's sign; Webspace tenderness test. Maximal ankle dorsiflexion and plantar percussion (MADAPP) test. Details of these tests can be found in appendix 5.
9. All participants will undergo a dynamic ultrasound scan of the affected area. Where a neuroma is identified by US, the location and size of the lesion will be recorded. In instances of multiple neuromas, either bilaterally or unilaterally, only the neuroma at the site of the participant's greatest discomfort shall be recorded. However, in order to limit the impact of the additional neuromas on pain scores and QoL scores, all neuromas will be treated. Where the US scan is negative for a neuroma the participant shall be removed from the study and invited to attend the QMU MSK clinic for further treatment. If the US scan identifies any other anomaly except a neuroma, the participant will be informed, withdrawn from the study and referred for the appropriate treatment.
10. Each participant shall be measured on the HR Walkway in order to assess forefoot loading patterns. The walkway mat will be set to obtain plantar pressure distribution measurements and will be set up in such a manner as to ensure that none of the systems cabling can interfere with the recording of each participant. Connecting the handle unit to the walkway sensor should change the status from "misaligned" to "sensor OK". The sensor handle units will be held in place by Velcro strips to ensure their placing is secure. The participant will be asked to walk along the mat for at least twenty steps in order to accomplish the "break in", after which, the computer will give live pressure readings from the sensors. Data acquisition parameters will include duration, frames to record, frequency and period. Once all parameters are set, data recording will commence. Participants will be asked to walk the full length of the marked out walkway at their normal walking pace. This will be repeated and recorded three times.
11. At this point all participants shall complete their second set of VAS scores and QoL questionnaires. This will be done on the same day as the first set but after the US scan and HR Walkway has been completed. This is to ensure that the VAS and QoL measurement tools are sufficiently robust, valid and repeatable. Allowing a time lapse with no therapeutic intervention should result in similar scores being obtained on both occasions, thereby inferring that the tools are measuring accurately.
12. All subjects will have their first pressure threshold meter (PTM) score recorded. This will be done by taking measurements of the metatarsophalangeal joint (MTPJ) either side of the affected webspace and using the lowest scoring joint for this and all subsequent measurements. Where there is ambiguity regarding the webspace, all lesser MTPJs will be measured and the lowest scoring joint used for all subsequent measurements. The PTM measurement will be taken in such a way that the readout display of the meter is covered so that it cannot be read. This will double blind the measurement so that neither the subject not the practitioner will have sight of the PTM measurement results until the intervention is complete.
13. Minimisation with weighted randomisation will be used to split subjects into two trial groups.
14. Those randomised to the steroid group shall receive a single injection of 1 mL methylprednisolone [40 mg] and 1 mL 2% lignocaine. They shall then be asked to return for review in six weeks. A second injection may be offered at this point if clinically indicated.
15. Those in the manipulation group shall have the lesser MTPJs of the affected foot manually manipulated using a high velocity, low amplitude thrust technique. They will be asked to return once each week for a further five weeks. At each visit the VAS and PTM measurements shall be repeated, as will the manual manipulation. They shall also be asked to return for a review in the sixth week.
16. All subjects will receive a weekly text message asking them to rate their pain on a scale of 0 - 10.
17. At the six week review the ultrasound scan, high resolution walkway, clinical tests, QoL questionnaires, VAS and PTM scores shall all be repeated. Subjects will then be asked to attend for a second review at three months.
18. The three month review shall follow the format of the six week review and subjects will be asked to attend for a six month and one year review where the same procedure shall be followed again.
19. At the end of the study, all data shall be processed and subject to statistical analysis. Comparisons will be drawn between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria shall be any positive clinical sign together with a positive diagnostic ultrasound giving rise to a diagnosis of Morton's neuroma/plantar digital neuritis.
* A VAS score of no less than 25/100 will also be required.
* All subjects must be over 18 years of age and able to offer informed consent.

Exclusion Criteria:

* Absolute exclusion criteria will include Rheumatoid Arthritis, recent (less than 3 months) fracture to the affected foot, peripheral neuropathy, localised infection, pregnancy, allergy to Methylprednisolone.
* Allergy to local anaesthetic.
* Further exclusion criteria include Active infection
* Diabetes mellitus
* Ulcerative colitis
* Diverticulitis
* Hypothyroidism
* Osteoporosis
* Renal impairment
* Hepatic impairment and Coagulation disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Visual analogue pain scale | baseline then every 3 months until one year after randomisation
  Assessing change from baseline to one year in recorded visual analogue pain scales

SECONDARY OUTCOMES:
Algometric pressure threshold testing | every 3 months until one year after randomisation
  Assessing change from baseline to one year in recorded Algometric pressure threshold scores
Manchester - Oxford Foot Questionnaire | every 3 months until one year after randomisation
  Assessing change from baseline to one year in recorded Manchester - Oxford Foot Questionnaire scores
The Foot and Ankle Ability Measure | every 3 months until one year after randomisation
  Assessing change from baseline to one year in recorded The Foot and Ankle Ability Measurements
SF-36 Questionnaire | every 3 months until one year after randomisation
  Assessing change from baseline to one year in recorded SF-36 Questionnaire scores

CONTACTS AND LOCATIONS:
Overall Officials: Derek Santos, PhD, Study Director — Queen Margaret University
Locations (1):
- Queen Margaret University, Musselburgh, Lothian, United Kingdom